CLINICAL TRIAL: NCT01570582
Title: A Phase II Randomized Controlled Clinical Trial of Carboplatin and Paclitaxel or Carboplatin and Gemcitabine in Platinum-sensitive, Recurrent Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Brief Title: A Phase IIclinical Trial of Carboplatin and Paclitaxel or Carboplatin and Gemcitabine in Platinum-sensitive, Recurrent Ovarian, Fallopian Tube, and Primary Peritoneal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Korean Gynecologic Oncology Group (Other)
Responsible Party: Principal Investigator, Taek Sang Lee, Principal Investigator, Korean Gynecologic Oncology Group
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KGOG3017
Record Dates: First submitted 2012-03-14; First posted 2012-04-04 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cancer
Keywords: recurrent ovarian; ECG; GOG performance; Hematologic g; Blood chemistry and urinalysis h
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Carboplatin; Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- drug effect (Experimental): Subjects assigned to Arm I Neople taksoljuwa Latin week the first day of the week based outpatient / inpatient treatment receive it. The subjects first received taksoljureul given over 3 hours followed by 30 minutes will be administered Neople Latin week.
  Subjects assigned to Arm II Gemcitabine and Latin Neople every week based on the first day of the outpatient / inpatient treatment receive it. The subjects first received Gemcitabine given over 30 minutes followed by 30 minutes will be administered Neople Latin week.
  Gemcitabine and eighth day of the foreign / hospitalization are given over 30 minutes.
  Regimen of the progression of the disease, the subject can not continue to deny or toxic dose every 3 weeks until at least 6 cycles should be administered to. Subjects completed six cycles of medication which responds subjects, the researchers believe it is necessary to sustain if the regimen is
  Interventions: Drug: carboplatin and paclitaxel

INTERVENTIONS:
Drug: carboplatin and paclitaxel — Subjects assigned to Arm I Neople taksoljuwa Latin week the first day of the week based outpatient / inpatient treatment receive it. The subjects first received taksoljureul given over 3 hours followed by 30 minutes will be administered Neople Latin week.
  Other Names: carboplatin , paclitaxel and Gemcitabine

SUMMARY:
purpose Primary endpoint

* To evaluate the 24 month disease free survival Second endpoints
* To evaluate the 24 month overall survival To analyze the toxicity and the quality of life

DETAILED DESCRIPTION:
Approximately 48 month from the date of IRB approval

Patients enrolled in this study targets approximately 314 people. Completion of patient enrollment is expected to take approximately 24 month, approximately 24 month follow-up period is expected to be needed

ELIGIBILITY:
Inclusion Criteria:

* Patients with epithelial ovarian, fallopian tube cancer bokmakam or pathological diagnosis of recurrent states there must be must be present.
* Pathologically Serous adenocarcinoma, endometrioid adenocarcinoma, mucinous adenocarcinoma, undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, transitional cell carcinoma, malignant Brenner's Tumor, or adenocarcinoma not otherwise specified (NOS) have been diagnosed with possible participation.
* Patients with CA-125 (biochemical recurrence), as described below elevation or clinically measurable lesions or the measurement is not possible, as there should be evidence of recurrence.
* If at least one (record as the longest diameter) can be accurately measured in at least one lesion that is defined. For each lesion, such as MRI or CT, when measured by traditional methods should be at least 20mm spiral CT (spiral CT) have been measured to be less than 10mm when.
* Neutrophil (ANC) by 1500 / ㎣ more Platelet count 100,000 / ㎣ more Serum creatinine concentration 1.5mg/dL (133mol / l) or creatinine clearance less than 60ml/min should be at least two.

Exclusion Criteria:

* Patients must be at least 18 years of age.
* Patients with epithelial ovarian, fallopian tube cancer bokmakam or pathological diagnosis of recurrent states there must be must be present.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2010-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
24month progression free survival | 24 months

SECONDARY OUTCOMES:
Toxicity Profile | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Korea Institute of Radiological and Medical Sciences, Seoul, South Korea